CLINICAL TRIAL: NCT02378428
Title: A Phase II Study of <131>I-Metaiodobenzyguanidine (<131>I-MIBG) Therapy for Patients With MIBG Avid Tumors
Brief Title: MIBG Therapy for Patients With MIBG Avid Tumors
Acronym: MIBG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-00656; NCH MIBG (Other: Columbus CRI)
Record Dates: First submitted 2014-03-04; First posted 2015-03-04 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: MIBG Avid Tumors
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MIBG (Experimental): Research participants with MIBG avid tumors
  Interventions: Drug: MIBG

INTERVENTIONS:
Drug: MIBG
  Other Names: <131>I-Metaiodobenzylguanidine

SUMMARY:
This is a Phase II study for patients with MIBG avid tumors. The study is to determine the response rate to <131>I-MIBG in patients with de novo, relapsed or refractory neuroblastoma or other MIBG avid malignant tumors 42 days post MIBG therapy. It will also be evaluating the tolerability and safety of the study agent by evaluating the hematopoietic and non-hematopoietic toxicity of <131>I-MIBG therapy. Tumor response will be evaluated by comparing the patient's disease pre-treatment against the patient's day +42 post <131>I-MIBG treatment. The evaluations may include the following: <131>I-MIBG scan, CT or MRI, urine catecholamine, bone marrow analyses and any other tests considered standard of care for cancer evaluation. To be eligible for participation, patients must have tumors that are MIBG avid. Patients must also have a stem cell source for autologous rescue in the event of protracted therapy associated cytopenias. Peripheral stem cell collections are preferred as the hematopoietic cell source. Bone marrow harvests for a hematopoietic cell source is an alternative. This study will provide data for future clinical trials utilizing <131>I-MIBG therapies. A room on H12 has been prepared with lead lined walls, and many radiation safety components to accomodate this treatment. <131>I metaiodobenzlguanidine (<131>I-MIBG) is a radiopharmaceutical that concentrates within adrenomedullary tissue. The agent was initially used for tumor imaging due to its capability to locate pheochromocytomas, neuroblastomas and other neuroendocrine tumors. <131>I-MIBG was subsequently used as an therapeutic agent for these tumor types. Phase I and II therapeutic trials targeting neuroblastoma have reported response rates of 10-50%. Toxicities observed have been mainly hematopoietic, with ~50% of patients receiving 15mCi/kg requiring stem cell reinfusion. Observed non-hematopoietic toxicities have been mild. Most recently, trials have been conducted combining the study agent with myeloablative chemotherapy and stem cell reinfusion have been performed with initial response rates of ~50%.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 12 months and 65 years at the time of enrollment
* Diagnosis: diagnosis of neuroblastoma or at the time of relapse by histology and/or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites
* Disease Status:

  1. The presence of refractory or progressive disease (PD)
  2. For patients with neuroblastoma, the presence of mixed response (MR), or no response (NR) following the completion of A3973 or equivalent induction therapy, or the presence of a partial response (PR) with high Curie score (>2) following induction therapy.
  3. Patients with de novo high risk neuroblastoma who have completed standard induction therapy and do not achieve a CR, VGPR, or PR with low Curie score post induction.

     * Patients must have evidence of MIBG avid disease as determined by diagnostic MIBG scan obtained within 4 weeks of study entry.
* Patients who receive greater than 12 mCi/kg are required to have stem cell rescue products harvested prior to study treatment.
* Performance Level and Life Expectancy: Patients must have a Lansky Play Scale17 of 60% (<16 yrs old), Karnofsky score 60% (>16 yrs old), or ECOG score of < or equal to 2 and a life expectancy of 2 months.
* Patients may enter this study with or without salvage therapy for recurrent tumor. Patients must have fully recovered from the toxic effects of any prior therapy.
* Organ Function requirements:

Hematopoietic Criteria:

1. Hemoglobin- 10 gl/dl (transfusion allowed)
2. ANC- 550 / cu mm (off myeloid growth factors)
3. Platelets- > 50,000/cu mm. (transfusion allowed - however patients must not require more than two platelet transfusions per week).

Renal Function:

a. Serum Creatinine- < 2 x ULN for age.

Hepatic Function:

Total bilirubin <1.5 x ULN for age SGPT (ALT) and SGOT (AST) < 10 x ULN for age

Cardiac Function:

For children with NBL: Normal ejection fraction (>55%) documented by echocardiogram or radionuclide MUGA evaluation OR normal fractional shortening (>27%) documented by echocardiogram.

For subjects with paraganglioma/ pheochromocytoma: No clinically significant cardiac dysfunction.

Pulmonary Function:

Patients must have clinically normal lung function as manifested by no dyspnea at rest and no oxygen requirement

Reproductive Function:

1. Females of childbearing potential must have a negative pregnancy test within 1 week prior to treatment with 131I-MIBG.
2. Patients of childbearing potential must agree to use an effective birth control method.
3. Female patients who are lactating must agree to stop breast feeding

Exclusion Criteria:

* Pregnancy or breast feeding
* Have undergone a prior allogeneic BMT.
* Patients with disease of any major organ system that would compromise their ability to withstand therapy. Any significant organ impairment should be discussed with the Study Chair prior to patient entry.
* Patients who are on hemodialysis.
* Hepatitis B surface antigen (+) or Hepatitis C positive in preceding six months.
* Patients with an active infection requiring intravenous antivirals, antibiotics or antifungals. Patients on prolonged antifungal therapy are still eligible if they are culture negative and biopsy negative in suspected residual radiographic lesions have stabilized or regressed and they meet other organ function criteria.
* Prior total body irradiation, prior total abdominal or whole liver radiation
* Any medical or psychological condition or situation deemed by the PI to put the patient at increased risk of complications or noncompliance.
* Patients with curative treatment options.
* Patients for whom busulfan/ melphalan consolidation therapy following treatment with 131I-MIBG is planned.
* Patients for who CEM (carboplatin, etoposide, melphalan) therapy is administered within 30 days prior to 131I-MIBG therapy or for whom this therapy is planned within 30 days following administration of 131I-MIBG.

Ages: 12 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-03-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the response rate to <131>I-MIBG treatment. | Response rate will be assessed at 42 days post therapy.
  Responses will be defined by comparison to baseline studies obtained prior to study therapy. Disease status will be evaluated using CT/MRI scans, MIBG scans, plain films, as well as bone marrow aspiration and biopsy as dictated by the primary malignant diagnosis. Imaging modalities should be the same for pre and post MIBG assessments to facilitate response determination.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Ranalli, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States